CLINICAL TRIAL: NCT05495308
Title: Oncologic Results and Risk Factors for Recurrence in Patients With Locally Advanced Rectal Cancer and pCR After Neoadjuvant Treatment.
Brief Title: "Oncologic Results and Risk Factors for Recurrence in Patients With Locally Advanced Rectal Cancer and Pathologic Complete Response After Neoadjuvant Treatment. Results From an Observational Retrospective Multicenter Long-term Follow-up Study".
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Carlos Cerdán Santacruz, Colorectal Surgery Department at Hospital Universitario de la Princesa, Madrid. Spain. ORCID: 0000-0002-6507-900X, Hospital San Carlos, Madrid
Other Study IDs: C.I. 20/741-E
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer, Adenocarcinoma; Rectal Cancer Stage II; Rectal Cancer Stage III; Distant Metastasis; Local Recurrence of Malignant Tumor of Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 80 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NON-DISTANT METASTASES: Those patiens who do not develop distant metastasis during the follow-up time.
  Interventions: Procedure: neoadjuvant treatment
- DISTANT METASTASES: Those patiens who develop distant metastasis during the follow-up time.
  Interventions: Procedure: neoadjuvant treatment

INTERVENTIONS:
Procedure: neoadjuvant treatment — We study the number of patients who achive a complete pathological response after neoadjuvant treatment with radiochemotherapy.

SUMMARY:
Pathologic complete response (pCR) after multimodal treatment for locally advanced rectal cancer (LARC) patients is considered as the gold-standard of treatment success as it is associated to privileged oncologic outcome. Nevertheless, data from multicenter high-volume cohorts with long term follow-up are scarce.

This is a multicenter observational study using prospectively collected data from the Spanish Rectal Cancer Project database.

The main objective of the study is to update long-term oncologic follow-up of those patients treated for LARC with nCRT and surgery (either TME or subtotal TME; S-TME) who had obtained a pCR.

Secondary objective is to analyze demographic, clinical, operative and treatment variables in search of related factors to adverse oncologic outcomes, like distant recurrence or tumor-related deaths.

The results are reported in accordance with the STROBE (STrengthening the Reporting of OBservational studies in Epidemiology) Statement for observational studies.

All calculations are performed using Stata 13.1 (StataCorp, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological confirmation of rectal cancer preoperatively, in any of its histological variants.
* Tumor located less than 12 cm from the anal margin.
* Radiological stage II or III (cT3-4 N0 and/or any T with positive cN).
* Neoadjuvant treatment with radio-chemotherapy.
* Radical surgery performed on a scheduled basis and with curative intent.
* Definitive pathology study with complete tumor regression.

Exclusion Criteria:

* Patients operated on with palliative intent.
* Patients diagnosed with a hereditary colorectal cancer syndrome.
* Patients who presented synchronous metastases at the time of diagnosis, or concurrent malignancy of another origin.
* Patients who underwent emergency surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for LARC with nCRT and surgery (either TME or subtotal TME; S-TME) who had obtained a pCR
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to update long-term oncologic follow-up of those patients treated for LARC with nCRT and surgery (either TME or subtotal TME; S-TME) who had obtained a pCR. | May 2022-June 2022
  Patients treated for LARC with nCRT and surgery (either TME or subtotal TME; S-TME) who had obtained a pCR.

SECONDARY OUTCOMES:
To analyze operative and treatment data in search of related factors to adverse oncologic outcomes, like distant recurrence or tumor-related deaths. | May 2022-June 2022
  Operative and treatment data related to adverse oncologic outcomes.
To analyze demographic data in search of related factors to adverse oncologic outcomes, like distant recurrence or tumor-related deaths. | May 2022-June 2022
  Age (years) related to worse long-term oncologic outcomes.
To analyze further demographic data in search of related factors to adverse oncologic outcomes, like distant recurrence or tumor-related deaths. | May 2022-June 2022
  Normal Pretreatment CEA (ng/dl) related to worse long-term oncologic outcomes.
To analyze clinical data in search of related factors to adverse oncologic outcomes, like distant recurrence or tumor-related deaths. | May 2022-June 2022
  Tumour location (cm) and Distance from anal verge (cm) related to worse long-term oncologic outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided